CLINICAL TRIAL: NCT05258331
Title: An Open-label, Dose-escalation, Phase 1 Trial to Investigate the Safety, Tolerability, and Efficacy After Single- and Multiple-dose Administration of CT303 in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: Clinical Trial to Evaluate the Safety, Tolerability and Efficacy of CT303 in Patients With Psoriasis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: GC Cell Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT303A101
Record Dates: First submitted 2022-02-14; First posted 2022-02-28 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-02

CONDITIONS: Moderate to Severe Plaque Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): CT303
  Interventions: Genetic: CT303

INTERVENTIONS:
Genetic: CT303 — 1. Cohort 1 : Single-dose administration, intravenous injection
     * Dose 1(Starting dose) : 1.0*10^6 cells/kg
     * Dose 2 : 2.0*10^6 cells/kg
     * Dose 3 : 3.0*10^6 cells/kg
  2. Cohort 2 : Multiple-dose administration, intravenous injections (Week 0, Week 4)
     * Dose 1(Starting dose) : 1.0*10^6 cells/kg
     * Dose 2 : 2.0*10^6 cells/kg
     * Dose 3 : 3.0*10^6 cells/kg

SUMMARY:
Investigate the Safety, Tolerability, Efficacy and pharmacodynamics properties of CT303 in patients with moderate to severe plaque psoriasis

DETAILED DESCRIPTION:
This study is a multi-center, open-label, dose-escalation and dose-finding phase 1 clinical trial. The primary purpose is to evaluate the safety and tolerability of CT303 and the secondary purpose is to evaluate the safety and efficacy of CT303 in patients with moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 19 years old
2. Plaque psoriasis diagnosed before ≥ 6 months who did not show a sufficient response to one or more of the traditional systemic treatments or require change of treatment due to intolerance
3. Have moderate to severe plaque psoriasis as defined by PASI score ≥ 12, BSA ≥ 10% and sPGA score ≥ 3
4. Patients who have voluntarily decided to participate in the study and signed the informed consent form

Exclusion Criteria:

1. Guttate psoriasis, erythrodermic psoriasis, palmoplantar psoriasis, drug-induced psoriasis, and inverse psoriasis
2. History of treatment with cell therapy products including but not limited to mesenchymal stem cells
3. Have hypersensitivity, or medical history of clinically significant hypersensitivity, to the IP or its excipients
4. Current or history of cardiovascular diseases
5. Clinically significant hemorrhagic diseases, or gastrointestinal, respiratory, endocrinal, musculoskeletal, or neuropsychiatric disorders that are deemed by the investigator to be a potential threat to the safety of the subject due to study participation
6. Use of anticoagulants within 7 days prior to IP administration
7. Following treatment history for psoriasis

   * Use of topical therapy within the past 2 weeks
   * Use of phototherapy and/or systemic therapy within the past 4 weeks
   * Use of biologics within the past 4 to 24 weeks
8. Severe infection or other uncontrolled active infectious diseases requiring administration of systemic antibiotics, antivirals, etc. within 4 weeks prior to IP administration
9. Systemic or local inflammatory diseases requiring systemic anti-inflammatory treatment within 4 weeks prior to IP administration
10. Received or are scheduled to receive a live/live attenuated viral/bacterial vaccination within 12 weeks prior to IP administration (within 12 months for BCG vaccines)
11. Require administration of any prohibited concomitant medication specified in this protocol during participation in the study
12. QTc interval > 480 msec
13. Any of the following abnormalities or abnormal findings from laboratory tests:

    * AST or ALT > 3 times the upper limit of normal
    * Serum creatinine > 1.5 times the upper limit of normal
    * ANC < 1,500/μL, Hemoglobin < 10 g/dL, Platelet count < 100,000/μL
14. Hepatitis B or C infection or positive test for HIV at screening
15. History of malignant tumors within the last 5 years prior
16. Received or used any other IP or investigational device within 4 weeks prior to IP administration
17. Pregnant or breast-feeding women, or women of childbearing potential and men who do not agree to abstinence or use of effective methods of contraception from the time of obtaining informed consent and during the study
18. Patients who are deemed ineligible to participate in the study for other reasons by the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
TEAE (treatment-emergent adverse event) incidence rate | Day 0 to Day 28
  Evaluate safety through the incidence rate of TEAE (treatment-emergent adverse event) after CT303 administration

CONTACTS AND LOCATIONS:
Overall Officials: Seongjin Jo, Principal Investigator — Seoul National University Hospital
Locations (3):
- South Korea (3):
  - CHA Medical School Bundang CHA Medical Center, Gyeonggi-do
  - Pusan national university hospital, Pusan
  - Seoul national university hospital, Seoul

IPD SHARING:
Plan to Share IPD: No